CLINICAL TRIAL: NCT01771328
Title: Continuous Subcutaneous Hydrocortisone Infusion in Congenital Adrenal Hyperplasia
Acronym: CAH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2012/749
Record Dates: First submitted 2013-01-10; First posted 2013-01-18 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Adrenal Hyperplasia, Congenital
Keywords: Adrenal Hyperplasia, Congenital
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital | interventions — Hydrocortisone; hydrocortisone hemisuccinate; Cortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hydrocortisone (Active Comparator): Treatment B ( Solu-Cortef) the initial standard dose of 10mg/m2/24hrs. Hydrocortisone infusate will be given as Solu-Cortef Act-o-Vial 50mg/ml, produced by Pfizer. Treatment will take 4 months.
  Interventions: Drug: Hydrocortisone
- cortisone acetate (Active Comparator): Treatment A (Cortisone tbl.) is current treatment, i.e. glucocorticoid and mineralocorticoid replacement according to best clinical judgement. This treatment period will take 6 months.
  Interventions: Drug: Cortisone acetate

INTERVENTIONS:
Drug: Hydrocortisone — Initial standard dose of 10mg/m2/24hrs administered by pump during the treatment period, it will take 4 months. Body surface area will be calculated according to the nomogram from the formula of Du Bois and Du Bois.
  Other Names: Solu-Cortef
  Arms: hydrocortisone
Drug: Cortisone acetate — Patients will take this tables two times during day according to best clinical practice of therapy of congenital adrenal hyperplasia. Usually Cortisone 25 mg 1 tbl. in the morning and Cortisone 25 1/4 tbl. in the evening. This period will take 6 months.
  Other Names: Cortisone
  Arms: cortisone acetate

SUMMARY:
The conventional glucocorticoid replacement therapy in congenital adrenal hyperplasia (CAH) renders the cortisol levels unphysiological, which may cause symptoms and long-term complications. Glucocorticoid replacement is technically feasible by continuous subcutaneous hydrocortisone infusion (CSHI), and can mimic the normal diurnal cortisol rhythm. This method was recently applied to treat a patient through a critical phase of puberty. This is a clinical trial aiming to evaluate CSHI treatment in patients with CAH. The main objective is to determine the effects of CSHI on metabolic parameters (androstenedione and 17-hydroxyprogesterone profiles, and testosterone,adrenocorticotropic hormone(ACTH), cortisol, and bone markers), and to determine the required glucocorticoid doses. Secondary objectives are to determine effects on clinical status, body weight, blood pressure and other metabolic parameters, as well as on subjective health status (AddiQoL, SF36).

DETAILED DESCRIPTION:
CAH patients are treated with glucocorticoids and mineralocorticoids. Ideally, the glucocorticoid doses should be sufficient to suppress the elevated ACTH secretion, and hence attenuate the increase in androgen levels. Because of this, CAH patients use higher steroid doses than patients with autoimmune adrenal insufficiency (Addison's disease) and therefore are in higher risk of developing glucocorticoid side effects. The natural glucocorticoids, hydrocortisone (cortisol) or cortisone acetate, are preferred during childhood because of the growth suppressive effects of the longer acting synthetic glucocorticoids, prednisolone and dexamethasone. There is no consensus as to which type of glucocorticoid and which doses should be used for adult CAH patients. Glucocorticoids display a typical diurnal variation, which the current therapy does not restore, leading to both to over- or undertreatment. Some CAH patients experience symptoms that may be due to unphysiological glucocorticoid replacement therapy.

For selected CAH patients with poor response to conventional replacement therapy, or with problematic side effects such as impaired growth, weight gain, metabolic syndrome, and osteoporosis, continuous subcutaneous hydrocortisone infusion (CSHI) might become a treatment option. CSHI treatment would also be facilitated by the use of the small disposable pumps now developed for insulin treatment.

CSHI: Pharmacodynamics, Pharmacokinetics, and safety Hydrocortisone is identical to cortisol; the pharmacodynamics does not depend on mode of delivery. A hydrocortisone solution can be safely applied for three days in the insulin pump without major day-to-day variation. A daily dose of 10 mg/m2 body surface area/day restores normal levels of saliva cortisol in most patients. Thus, it is possible to mimic the physiological diurnal cortisol variation seen in healthy subjects.

The study will compare two glucocorticoid replacement modalities in randomised order within each patient. Prior to Baseline there will be a period of dose adjustment for pump treatment. Patients will be educated in groups, and dose adjustments will be co-ordinated with regular visits at the outpatient clinic/telephone consultation combined with laboratory analyses.

The patients will be assigned a participation number and randomised to any of two treatment sequences (A-B or B-A). Should the need for an extra glucocorticoid dose occur (intercurrent illness) during the study, the patients should administer their previous glucocorticoid replacement for safety reasons. Extra doses should be recorded in the patient diary. Treatment A is current treatment, i.e. glucocorticoid and mineralocorticoid replacement according to best clinical judgement. Treatment B is CSHI with the initial standard dose of 10mg/m2/24hrs. Body surface area will be calculated according to the nomogram from the formula of Du Bois and Du Bois.

After 7 days after initiating pump therapy the patient should be reassessed with blood dots (17-hydroxyprogesterone) and saliva cortisol and saliva 17-hydroxyprogesterone measurements in the morning (0800-0900) and in the evening (2300-2400). Based on results of this testing the dose will be changed at the discretion of the investigator. The further new testing should be done within 7-10 days.

When the final dose is established a 24h urine measurement, blood test in the morning (17-hydroxyprogesterone and cortisol) and a salivary sample full profile (full profile Hrs. 0800, 0930, 1100, 1230, 1700, 2100, 2400, 0300), will be done before entering the study. The dose adjustment period will be unlimited but will take minimally 4 weeks (aiming to obtain normal range levels of morning serum cortisol (160- 620 nmol/l), and 3-4 times increase in morning serum 17-hydroxyprogesterone (0,3-8,6 nmol/l for females, 0,9-6,6 nmo/l for males), and midnight (24:00) saliva cortisol (<2,8 nmol/l) and a circadian pattern as indicated in figure 1.

Afterwards it will 4 weeks wash out period before starting, wash out period between treatments modalities will take 2 months.

ELIGIBILITY:
Inclusion Criteria:

* verified salt-wasting CAH and simple virilizing CAH, on single prednisone, or hydrocortisone therapy.
* In case of concomitant endocrine/autoimmune diseases these should be on stable treatment during the study period.

Exclusion Criteria:

* Patients with diabetes mellitus on insulin pump treatment will not be included in this study
* cardiovascular disease, active malignant disease and pregnancy, and pharmacological treatment with glucocorticoids or drugs that interfere with cortisol metabolism (antiepileptics, rifampicin, St. Johns wart).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-02; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Androgen levels | 3 months
  Androgen levels as parameters of adequate suppression of androgen production

SECONDARY OUTCOMES:
Steroid metabolism | 4 months
  levels of ACTH
bone metabolism | 3 months
fasting glucose | 4 months
body mass index | 3 months
Dual-energy X-ray absorptiometry (DXA) | 6 months
  body composition, bone mineral density
Subjective health status | 3 months
  questionnaire
waist circumference | 3 month
  cm
hip circumference | 3 months
  cm
blood pressure | 3 months
fasting insulin | 3-4 months
glycated haemoglobin (Hb1AC) | 4 months
lipid levels | 4 months
c-reactive protein | 4 months
Steroid metabolism | 4 months
  cortisol levels

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Løvås, MD, PhD, Principal Investigator — Haukeland University Hospital, Department of Medicine
Locations (1):
- Haukeland Universitetssykehus, Department of Medicine, Bergen, Norway

REFERENCES:
- See also: Related Info — http://www.ese-hormones.org/